CLINICAL TRIAL: NCT02675998
Title: An 8-week, Multicenter, Randomized, Double-Blind, Parallel Group Study With a 4-week, Placebo-Controlled, Randomized Withdrawal Period to Evaluate the Efficacy, Safety, and Tolerability of Tenapanor to Treat Hyperphosphatemia in End-Stage Renal Disease Patients on Hemodialysis (ESRD-HD)
Brief Title: An 8-Week Study to Evaluate Tenapanor in the Treatment of Hyperphosphatemia in End-Stage Renal Disease Patients on Hemodialysis (ESRD-HD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TEN-02-201
Record Dates: First submitted 2016-02-03; First posted 2016-02-05 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — tenapanor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 3mg BID (Experimental): Tenapanor, 3mg BID (6mg total)
  Interventions: Drug: Tenapanor
- 10mg BID (Experimental): Tenapanor, 10mg BID (20mg total)
  Interventions: Drug: Tenapanor
- Dose Titration (Experimental): Tenapanor, patients start at 30mg BID and can down titrate weekly to 20, 15, 10, and 3mg BID, sequentially based on a GI tolerability question
  Interventions: Drug: Tenapanor
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenapanor
  Other Names: RDX5791, AZD1722
  Arms: 10mg BID; 3mg BID; Dose Titration
Drug: Placebo
  Arms: Placebo

SUMMARY:
This phase 3, 8-week, randomized, double-blind, parallel group, multi-center study with a 4-week, placebo-controlled, randomized withdrawal period will evaluate the efficacy, safety and tolerability of Tenapanor to treat hyperphosphatemia in end-stage renal disease patients on hemodialysis (ESRD-HD). Subjects who qualify are randomized into the study will either receive 3 mg BID, 10 mg BID, or a titration regimen of tenapanor.

DETAILED DESCRIPTION:
The study consists of a screening visit, a wash out period of up to 3 weeks, when existing phosphate lowering medication is withheld, an 8-week treatment period, in which all groups receive tenapanor, and a 4-week placebo-controlled, randomized withdrawal period, during which patients are re-randomized 1:1 to either remain on their current tenapanor treatment or placebo.

Depending on the increase in serum phosphate levels, subjects can be randomized 1,2, or 3 weeks after being taken off their phosphate lowering medication.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* Females must be non-pregnant, non-lactating, and either be post-menopausal for at least 12 months, have documentation of irreversible surgical sterilization, or confirm the use of one of the acceptable contraceptive methods.
* Males must agree to avoid fathering a child and agree to use an appropriate method of contraception
* Chronic maintenance hemodialysis 3x/week for at least 3 months
* Kt/V ≥ 1.3 at most recent measurement prior to screening
* Prescribed and taking at least 3 doses of phosphate binder per day
* Serum phosphate levels should be between 4.0 and 7.0 mg/dL (inclusive) at screening
* For randomization in the study, after 1 week wash-out of phosphate binders, subjects must have serum phosphate level of at least 9 mg/dL but below 10 mg/dL and have had an increase of at least 1.5 mg/dL versus pre-wash out value
* For randomization in the study, after 2 or 3 weeks wash-out of phosphate binders, subjects must have serum phosphate level of at least 6 mg/dL but below 10 mg/dL and have had an increase of at least 1.5 mg/dL versus pre-wash out value

Exclusion Criteria:

* Severe hyperphosphatemia defined as >10 mg/dL on Phosphate-binders at any time point during clinical routine monitoring for the 3 preceding months before screening
* Serum parathyroid hormone >1200 pg/mL
* Persistent metabolic acidosis defined as serum carbon dioxide <18 mmol/L from two consecutive measurements during screening and washout periods
* Clinical signs of hypovolemia at randomization
* History of inflammatory bowel disease (IBD) or diarrhea predominant irritable bowel syndrome (IBS-D)
* Scheduled for living donor kidney transplant, change to peritoneal dialysis, home HD or plans to relocate to another center during the study period
* Diarrhea or loose stools during the week before randomization defined as BSFS ≥ 6 and frequency ≥ 3 for 2 or more days
* Any evidence of or treatment of malignancy within one year, excluding non-melanomatous malignancies of the skin
* Positive serology with evidence of significant hepatic impairment or WBC elevation according to the Investigator
* Life expectancy < 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2018-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, Ph.D., Study Chair — Ardelyx, Inc.
Locations (32):
- United States (32):
  - Ardelyx Investigative Site 429, Huntsville, Alabama
  - Ardelyx Investigative Site 425, Riverside, California
  - Ardelyx Clinical Site 403, Denver, Colorado
  - Ardelyx Investigative Site 410, Lauderdale Lakes, Florida
  - Ardelyx Investigative Site 430, Miami, Florida
  - Ardelyx Investigative Site 427, Meridian, Idaho
  - Ardelyx Investigative Site 432, Shreveport, Louisiana
  - Ardelyx Investigative Site 415, Bethesda, Maryland
  - Ardelyx Investigative Site 402, Kalamazoo, Michigan
  - Ardelyx Investigative Site 424, Roseville, Michigan
  - Ardelyx Investigative Site 409, Brookhaven, Mississippi
  - Ardelyx Investigative Site 417, Columbus, Mississippi
  - Ardelyx Investigative Site 431, Tupelo, Mississippi
  - Ardelyx Investigative Site 423, St Louis, Missouri
  - Ardelyx Investigative Site 416, Albuquerque, New Mexico
  - Ardelyx Investigative Site 419, The Bronx, New York
  - Ardelyx Investigative Site 408, Asheville, North Carolina
  - Ardelyx Investigative Site 411, Charlotte, North Carolina
  - Ardelyx Investigative Site 420, New Bern, North Carolina
  - Ardelyx Investigative Site 426, Raleigh, North Carolina
  - Ardelyx Investigative Site 412, Wilmington, North Carolina
  - Ardelyx Investigative Site 414, Bethlehem, Pennsylvania
  - Ardelyx Investigative Site 404, Columbia, South Carolina
  - Ardelyx Investigative Site 421, Orangeburg, South Carolina
  - Ardelyx Investigative Site 428, Sumter, South Carolina
  - Ardelyx Investigative Site 413, Knoxville, Tennessee
  - Ardelyx Investigative Site 418, Nashville, Tennessee
  - Ardelyx Investigative Site 406, Austin, Texas
  - Ardelyx Investigative Site 405, Bellville, Texas
  - Ardelyx Investigative Site 422, San Antonio, Texas
  - Ardelyx Investigative Site 407, San Antonio, Texas
  - Ardelyx Investigative Site 401, St. George, Utah

REFERENCES:
- [Derived] Sprague SM, Weiner DE, Tietjen DP, Pergola PE, Fishbane S, Block GA, Silva AL, Fadem SZ, Lynn RI, Fadda G, Pagliaro L, Zhao S, Edelstein S, Spiegel DM, Rosenbaum DP. Tenapanor as Therapy for Hyperphosphatemia in Maintenance Dialysis Patients: Results from the OPTIMIZE Study. Kidney360. 2024 May 1;5(5):732-742. doi: 10.34067/KID.0000000000000387. Epub 2024 Feb 7. PMID 38323855
- [Derived] Silva AL, Chertow GM, Hernandez GT, Lynn RI, Tietjen DP, Rosenbaum DP, Yang Y, Edelstein S. Tenapanor Improves Long-Term Control of Hyperphosphatemia in Patients Receiving Maintenance Dialysis: the NORMALIZE Study. Kidney360. 2023 Nov 1;4(11):1580-1589. doi: 10.34067/KID.0000000000000280. Epub 2023 Oct 19. PMID 37853560

RESULTS

PARTICIPANT FLOW:
Groups:
- 3mg BID: Tenapanor, 3mg BID (6mg total)
  Tenapanor
- 10mg BID: Tenapanor, 10mg BID (20mg total)
  Tenapanor
- 30 mg Dose Titration: Tenapanor, patients start at 30mg BID and can down titrate weekly to 20, 15, 10, and 3mg BID, sequentially based on a GI tolerability question
  Tenapanor
- Randomized Withdrawal Period Placebo: These were participants re-randomized to placebo during the 4-week withdrawal period.
Period: 8-Week Treatment Period
Arm/Group | 3mg BID | 10mg BID | 30 mg Dose Titration | Randomized Withdrawal Period Placebo
Started | 74 | 73 | 72 | 0
Completed | 57 | 54 | 53 | 0
Not Completed | 17 | 19 | 19 | 0
Not completed — Adverse Event | 6 | 5 | 6 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 3 | 0
Not completed — Lack of Efficacy | 2 | 5 | 3 | 0
Not completed — Physician Decision | 1 | 0 | 2 | 0
Not completed — GI side Effects | 1 | 4 | 2 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 0
Not completed — Other | 3 | 1 | 2 | 0
Period: 4-Week Randomized Withdrawal Period
Arm/Group | 3mg BID | 10mg BID | 30 mg Dose Titration | Randomized Withdrawal Period Placebo
Started (The number of patients in combined tenapanor groups is less since half were re-randomized to Placebo) | 25 | 23 | 34 | 82
Completed | 24 | 22 | 32 | 74
Not Completed | 1 | 1 | 2 | 8
Not completed — Lack of Efficacy | 0 | 1 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: This was a placebo-controlled randomized withdrawal study. All participants received drug during the first 8-weeks (no placebo) and then were randomized 1:1 to either remain on tenapanor dose or receive placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | 3mg BID | 10mg BID | Dose Titration | Placebo | Total
Number analyzed (Participants) | 74 | 73 | 72 | 0 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (11.49) | 57.4 (10.81) | 54.2 (10.87) |  | 55.8 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 39 | 24 |  | 91
  Male | 46 | 34 | 48 |  | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 19 |  | 40
  Not Hispanic or Latino | 61 | 65 | 53 |  | 179
  Unknown or Not Reported | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 |  | 2
  Asian | 2 | 0 | 0 |  | 2
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 1 |  | 4
  Black or African American | 40 | 45 | 40 |  | 125
  White | 30 | 25 | 31 |  | 86
  More than one race | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 0 |  | 0
Body Mass Index [Mean (Standard Deviation); unit: m/kg^2] | 32.5 (8.52) | 33.6 (8.50) | 33.4 (8.15) |  | 33.1 (8.37)

OUTCOME MEASURES:

1. Primary Outcome: Placebo Adjusted Change in Serum Phosphate During Randomized Withdrawal Period From Pooled Tenapanor Arms
Description: Serum phosphorus difference between placebo and tenapanor in the change from the end of the 8 week treatment period to the end of the randomized withdrawal period in Efficacy Analysis Set. The efficacy analysis was pre-defined to be a pooled analysis of all tenapanor treated patients with a minimum of a 1.2 mg/dL decrease in serum phosphorus during the 8-week treatment period
Time Frame: 4 weeks
Population: Patients who completed the first 8-weeks and had a minimum of a 1.2 mg/dL decrease in serum phosphorus were included in the analysis. Also, it was a pre-specificied pooled analysis where all the tenapanor treated patients were combined thus all patients are included in the 30 mg dose titration group.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 3mg BID | 10mg BID | 30 mg Dose Titration | Placebo
Number analyzed (Participants) | 0 | 0 | 43 | 37
mg/dL |  |  | 1.4 (0.23) | 0.6 (0.21)
Statistical Analysis 1: Comparison: 30 mg Dose Titration vs Placebo; Test type: Superiority; p = 0.01, ANCOVA

2. Secondary Outcome: Change in Serum Phosphate During 8-Week Treatment Period
Description: Serum phosphorus difference between baseline (end of washout period) to the end of the 8 week treatment period in ITT analysis set
Time Frame: Baseline and 8 weeks
Population: There was no placebo group during the 8-week treatment period.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 3mg BID | 10mg BID | 30 mg Dose Titration | Placebo
Number analyzed (Participants) | 74 | 73 | 72 | 0
mg/dL | -1.1 (0.17) | -1.1 (0.17) | -1.1 (0.18) |
Statistical Analysis 1: Comparison: 3mg BID; Test type: Superiority; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: 10mg BID; Test type: Superiority; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: 30 mg Dose Titration; Test type: Superiority; p < 0.001, ANCOVA

ADVERSE EVENTS:
Time Frame: 12 weeks. The first 8 weeks were tenapanor only and during the last 4 weeks half of the tenapanor-treated patients from the first 8 weeks were randomized to receive placebo
Description: There was no placebo during the first 8-weeks
Groups:
- 30 mg Dose Titration: Tenapanor, patients start at 30mg BID and can down titrate weekly to 20, 15, 10, and 3mg BID, sequentially based on a GI tolerability question
- Randomized Withdrawal Period Placebo: The 164 patients that ended the 8 week treatment period were re-randomized 1:1 to stay on tenapanor or receive placebo. The patients in this group were re-randomized to receive placebo for the last 4 weeks of the study
Arm/Group | 3mg BID | 10mg BID | 30 mg Dose Titration | Randomized Withdrawal Period Placebo
All-Cause Mortality (participants affected / at risk) | 1/74 | 0/73 | 0/72 | 0/82
Serious Adverse Events (participants affected / at risk) | 1/74 | 0/73 | 0/72 | 0/82
Other Adverse Events (participants affected / at risk) | 22/74 | 30/73 | 34/72 | 7/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3mg BID (N=74) | 10mg BID (N=73) | 30 mg Dose Titration (N=72) | Randomized Withdrawal Period Placebo (N=82)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3mg BID (N=74) | 10mg BID (N=73) | 30 mg Dose Titration (N=72) | Randomized Withdrawal Period Placebo (N=82)
Diarrhea (Gastrointestinal disorders) | 22 (22) | 30 (30) | 34 (34) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days